CLINICAL TRIAL: NCT04280406
Title: The Effect of Preoperative Antibiotics on Peri-implant Crestal Bone Remodelling and Postoperative Pain: A Randomized Controlled Trial
Brief Title: The Effect of Preoperative Antibiotics on Peri-implant Healing
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Principal Investigator, Robert Durand, Associate Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CERC-20-001-P
Record Dates: First submitted 2020-02-17; First posted 2020-02-21 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Dental Implant Failed
Keywords: dental implants; antibiotics; bone; pain
MeSH Terms: conditions — Pain | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: double-masked parallel arm randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Active Comparator): - 500mg of azithromycin one hour before implant placement
  Interventions: Drug: Azithromycin
- control (Placebo Comparator): - identical placebo one hour before implant placement
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Azithromycin — azithromycin 500mg one hour before implant placement
  Arms: Test
Drug: Placebo oral tablet — identical placebo one hour before implant placement
  Arms: control

SUMMARY:
Introduction: In order to minimize postoperative morbidity and failures of dental implant therapy, several antibiotic regimens have been proposed in the literature. However, the extensive use of antibiotics in health care has been debated due to the adverse effects and bacterial resistance. Furthermore, the impact of preoperative antibiotics on peri-implant bone level is still not clear.

Objectives: The primary objective of this study will be to assess whether giving preoperative antibiotics (azithromycin 500mg) after implant placement over 7 days will influence peri-implant crestal bone levels after 4 months in healthy patients undergoing platform-switched implant placement. The secondary objectives will be to evaluate postoperative pain severity, surgery-associated morbidities, and 1-year implant survival rate.

Methods: Fifty individuals will be recruited in a double-masked 2-arm randomized clinical trial. Participants in the intervention group will receive 500mg of azithromycin 1 hour before implant placement. Participants in the control group will take one placebo 1 hour preoperatively. The changes in mesial and distal crestal bone level (primary outcome) will be measured at baseline and 4-month follow-up using standardized periapical radiographs. Pain severity and surgery-associated morbidities (secondary outcomes) will be evaluated by clinical examinations and self-administered questionnaires. Implant survival rate will be assessed at the 1-year follow-up. Descriptive and bivariate analyses will be used to analyze the data. A P value ≤ 0.05 will be considered statistically significant.

Clinical relevance: This study will be the first placebo-controlled double-blinded randomized clinical trial studying the effect of preoperative azithromycin on radiographical, clinical and patient-based outcomes after implant surgery. This type of design will reduce as much as possible the risk of bias and increasing the quality of evidence. The results from this study might help provide guidelines for clinicians that will optimize implant survival rate while decreasing antibiotics exposure to patients undergoing straightforward implant surgery.

DETAILED DESCRIPTION:
Background

There have been many antibiotic regimens used to minimize the risks of infections and consequently, increasing the survival rate of dental implants. Initially, it was recommended to give antibiotics at least 1 hour before implant placement followed by daily doses for 10 days. A survey of private dental practices in UK found that there was a wide variation of antibiotic regimens: prophylactic, postoperative, and combination of both pre-and postoperative antibiotics. A recent survey showed that there is no consensus among oral and maxillofacial surgeons in the U.S. Consequently, in order to prevent the overuse of antibiotics and the potential emergence of drug-resistant bacteria, it would be advisable to find an optimal protocol including an antibiotic therapy with a minimal duration while the implant survival rate would remain unchanged. A recent systemic review reported that a single preoperative dose compared to no antibiotic or placebo decreased significantly implant failure. However, the included trials presented high and unclear risk of bias.Therefore, there is a need to carry out well controlled clinical trials that are placebo-controlled and include patient-based outcomes in order to increase the quality of evidence supporting the use of preoperative antibiotics to increase dental implant success.

More specifically, it was recommended by the latest Cochrane review that 2 g of amoxicillin, a commonly used penicillin antibiotic in dentistry, be prescribed before dental implant placement to prevent implant failure. However, allergies to penicillin and its derivatives have been reported by 8% of the U.S. population. Another limitation of penicillin antibiotics is their short half-life, which is about one hour. On the other hand, azithromycin has shown promising results as an adjunct to periodontal therapy and exhibits low toxicity, few side effects, excellent tissue penetration and a long half-life of about 68 hours. It has also anti-inflammatory properties. These characteristics make this antibiotic an interesting alternative to amoxicillin for allergic patients and could potentially demonstrate higher efficacy at preventing peri-implant bone remodeling after implant placement and decreasing postoperative complications.

Therefore, the primary objective of this study is to determine whether giving preoperative antibiotics to healthy patients undergoing straightforward platform-switched implant placement will significantly influence crestal bone loss around dental implants. The test group will receive one dosage of azithromycin before implant placement. The control group will receive an identical placebo preoperatively. Questionnaires for pain and interference with daily activities assessment will be distributed to participants and will be filled for the first postoperative week. Signs of postoperative morbidity will be recorded at 1 week following the surgery and both clinical and radiographic data will be collected at 4 months postoperative to assess the implants status. A radiographic and clinical follow-up will be done 1 year after the surgery.

Objectives and research hypothesis

Main objective : To determine whether giving preoperative azithromycin before implant placement will significantly influence crestal bone change around implants.

Secondary objectives :

1. To assess the patient's perception of the post-operative healing process.
2. To assess the surgeon's perception of the post-operative healing process.

Null hypothesis: The study's null hypothesis is that there is no difference in crestal bone loss around implants between azithromycin and the placebo.

Materials & Methods

Subjects in this randomized, double blind, placebo-controlled clinical trial will be divided in two groups: one group will receive 500 mg of azithromycin 1 h prior surgery; the second group will receive an identical placebo 1 h prior surgery.

Dental implant(s) (Astra Tech Implant EV System™, Dentsply Sirona Co., York, PA, USA) will be placed in a one stage procedure, without simultaneous bone grafting, and will be inserted either at Dr. Durand's practice (Le Groupe des Parodontistes, 2222 boul. René-Lévesque O., suite #200, Montreal, QC H3H 1R6, Canada) or at the implantology clinic of the Université de Montréal - Faculty of Dentistry (CRIP), Montreal, QC, Canada by one of two board-certified specialists and implant surgeons (minimum of 5 years of experience). All participants will be instructed to rinse with chlorhexidine gluconate 0.12% for 1 min. just before surgery and to take 600mg of ibuprofen and 500mg of acetaminophen. A third party will give an envelope to the patient containing the antibiotic or identical placebo to be taken preoperatively and the patient's study number so both the surgeon and the patient will be unaware of the antibiotic regimen. Subjects will be randomly distributed to one of the two study groups:

Test group: 500 mg of azithromycin taken 1 hour preoperatively; Control group: Identical placebo taken 1 hour preoperatively.

Randomization will be stratified by number of implants (one vs. more than one), using a block size of four. Randomization will be done by a statistician using a computer-generated sequence (SAS proc plan) and it will be sealed in consecutively numbered opaque envelopes. The subjects will receive from a research assistant the envelopes containing either the preoperative placebo or the antibiotic. All participants will have to take the antibiotic (or placebo) and analgesics (ibuprofen 600mg and acetaminophen 500mg) under the supervision of the research assistant. They will have to fill the questionnaires to evaluate their medical and socio-demographic status, as well as preoperative pain and anxiety levels using self-reported questionnaires and a 10-cm visual analog scale (VAS). Measures of asepsis will include the use of sterile drapes over the supine body of the patient. Screw-type, root-form, two-pieces rough surfaced dental implants will be placed using a standard surgical protocol, following the manufacturers' recommendations under local anesthesia. Mucoperiosteal flaps will be used to access underlying alveolar bone for all implant surgeries. The healing abutment will be inserted, and soft tissues will be sutured with interrupted sutures. A standardized periapical radiograph will be taken perpendicular to the crestal bone to assess the baseline crestal bone level on the mesial and distal aspects of the implant using a bite registration material (Blu-Mousse®, Parkell Inc., Edgewood, U.S.A.) adapted to a paralleling device (XCP film holding system, Dentsply Rinn, Elgin, U.S.A.) for each participant. The customized bite registration will be kept for each patient in a cool room in a locked cabinet with the participant study identification number for the subsequent 4 months and 1-year radiographic evaluations. The duration of the surgery and length of the incision will be recorded by the surgeon. The participants will be asked to refrain from performing mechanical plaque control in the surgical area and be advised to remain on a soft diet during the first postoperative week. They will be prescribed 600mg of ibuprofen to take as needed. They will also be prescribed an emergency analgesic (500mg acetaminophen) to take if needed and a 0.12% chlorhexidine gluconate rinse to use twice daily until the sutures are removed 1 week later. After receiving the standardized verbal and written post-operative instructions, participants will be given questionnaires to assess postoperative pain and interference with daily activities for the first postoperative week. The patient will be asked to keep a pain medication diary to keep track of the number of analgesics (ibuprofen and acetaminophen) taken for the first postoperative week. The patient will be asked to record his/her experience with the interference with their daily activities using a 10-cm VAS questionnaire with end points being "none" and "extremely much" and will have to attribute a numerical value to his/her pain intensity experienced using the Numerical Rating Scale (NRS-11), with 0 representing "no pain" and 10 "intolerable". The patient's pain experience will be assessed immediately before surgery and will also be assessed with the daily pain medication intake diary. Since anxiety has been positively associated with pain experience after surgery, VAS of Anxiety will be given to patients before and after surgery and at the 1-week follow-up. Daily activities will include their ability to chew foods they want to eat, to open their mouth wide, talk, sleep, go to school or work, carry on a regular social life and participate in their favorite recreational activities. The subjects will be asked to bring back to the research assistant the pain and daily interference questionnaires as well as the pain medication diary and the envelope and drug containers to ensure their compliance with the prescriptions. At the end of the first postoperative control appointment, one calibrated examiner (IA) unaware of the antibiotic prescribed will collect the daily diary, will ask the patient to quantify his/her anxiety using a VAS, and will evaluate swelling, bruising, pus exudate and wound dehiscence as described elsewhere. Postoperative swelling will be graded as follows: 0 = No swelling, 1 = Mild swelling, 2 = Moderate swelling, 3 = Severe swelling. Postoperative bruising, suppuration and wound dehiscence will be evaluated using Boolean variables: 0 = None; 1 = Present. The examiner will then measure the modified plaque index (PI) at four sites per implant (mesial, distal, buccal, lingual). The PI is graded as follows: 0 = no detection of plaque, 1 = Plaque only detected by running a probe (PCP-UNC15; Hu-Friedy Mfg Co., Chicago, U.S.A.) along the smooth surface of the healing abutment, 2 = Plaque can be seen by the naked eye, 3 = Abundance of soft matter. The PI will be also measured at the 16-weeks and 1-year examinations. At the 16-weeks evaluation, the implants will be re-assessed both clinically and radiographically to confirm osseointegration and the modified PI by an investigator. In addition, probing depth (PD) on 4 sites per implant and bleeding upon probing (BI index) will be measured. This appointment will coincide with the impression for restoration of the implant. The same calibrated examiner unaware of the antibiotic taken will verify if the implants are osseointegrated by taking a standardized periapical radiograph to verify the presence or absence of infection and evaluate crestal bone loss using the standardized bite registration and paralleling device. The examiner will also assess implant mobility using the handles of two blunt dental instruments (osseointegration = immobile, failure = mobile) and the presence or absence of any symptom related to infection (suppuration), inflammation (erythema, bleeding on probing) or neuropathy (paresthesia, dysesthesia, anesthesia). One year after the implant placement, a standardized radiograph will be taken to measure crestal bone loss. The PD and BI will be redone at the 1-year follow-up as well as presence or absence of infection assessment by the calibrated examiner. Crestal bone level changes (mm) will be measured on mesial and distal aspects of implants using superimposed images and a software (Adobe Ilustrator CC 2017 (Adobe systems Inc. San Jose, CA, U.S.A.) by one investigator who is unaware of the antibiotic regimen taken by the participants.

The primary outcome measures will be crestal bone loss at the mesial and distal aspects of each implant. The secondary outcomes will be the presence or absence of peri-implant radiolucency, patient's pain and anxiety experience (intensity (VAS) and number of analgesics taken), surgeon's perception of healing (intensity of swelling and presence/absence of bruising, pus exudate and wound dehiscence), modified PI, PD, BI, presence or absence of implant mobility, presence or absence of pain, infection, neuropathies, and presence or absence of pus exudate.

Statistical analysis

The trained and calibrated examiner will perform all clinical measurements and take the radiographs. An intra- and inter-reliability study will be done to compare with a gold standard examiner. One calibrated examiner will perform the radiographic analysis. Cohen's kappa, intraclass correlation coefficient and Bland and Altman graphs will be used to evaluate reliability. Normality of data distribution will be assessed using the Shapiro-Wilk test. Crestal bone loss, PD and patient's pain and anxiety perception (VAS) will be analyzed with repeated measures ANOVA or nonparametric ANOVA-type statistic, with time as a repeated measure (7 days) and groups as a between group measure. Groups will be compared regarding postoperative swelling with Mann-Whitney U test. Groups will be compared regarding implant survival at 4 months, bruising, suppuration, wound dehiscence, mobility, presence of pus exudate, PI, BI, presence of peri-implant radiolucency on the radiographs, and presence of persistent signs/symptoms with the Fisher's exact test. Analyses will be conducted in conformity of the intention to treat principles.

ELIGIBILITY:
Inclusion Criteria:

* Periodontally healthy remaining dentition or presenting with mild gingivitis with adequate oral hygiene.
* Presence of a partially edentulous alveolar ridge that is planned to be restored with no more than 2 implants.
* To have 1 or 2 implants restored with a crown or fixed bridge.
* Presence of a non-infected site.
* Presence of enough bone and soft tissue for the implant to be placed without additional bone augmentation in a 1-stage approach (with healing abutment).
* Implants 6 mm long or longer.
* Subjects able and willing to provide written informed consent and comply with study procedures.

Exclusion Criteria:

* Subjects taking regular analgesics or antidepressants.
* Smoking 10 cigarettes/cigars or more per day.
* Marijuana smokers.
* Use of vaping devices or e-cigarettes
* Drug abuse.
* Completely edentulous individuals.
* Pregnant and nursing women.
* Allergies to macrolides, and/or non-steroidal anti-inflammatory analgesics.
* Active peptic ulcers or susceptibility to peptic ulcers.
* Any systemic or local immunodeficiency.
* Any blood coagulation impairment or taking anticoagulants (ex.: Coumadin).
* Presence of uncontrolled periodontitis or poor oral hygiene.
* Presence of any acute oral infection.
* Presence of uncontrolled diabetes or other systemic diseases.
* Previous radiation therapy in the head and neck area.
* Intravenous bisphosphonates.
* Oral bisphosphonates intake for more than 4 years.
* Long-term intake of corticosteroids.
* Need for routine prophylactic antibiotics prior dental surgery.
* No intake of antibiotics 3 months prior surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
peri-implant crestal bone change | 4 months, 1 year
  variations in mm of the alveolar bone around each implant

SECONDARY OUTCOMES:
pain severity | preop and daily for 1 week
  postoperative visual analog scale pain assessment (10-cm line, 0 = no pain, 10 = worst pain ever)
interferences with daily activities | daily for 1 week
  postoperative visual analog scale assessment of interferences with daily activities (10-cm line, 0 = none, 10 = extremely much)
postoperative morbidities A | 1 week, 4 months, 1 year
  semi-quantitative assessment of flap dehiscence (0 = None; 1 = Present) at one week
postoperative morbidities B | 1 week, 4 months, 1 year
  semi-quantitative assessment of suppuration (0 = None; 1 = Present)
postoperative morbidities F | 4 months, 1 year
  pain (0 = None; 1 = Present) at 4 months and 1 year
postoperative morbidities G | 4 months, 1 year
  infection (0 = None; 1 = Present) at 4 months and 1 year
postoperative morbidities E | 4 months, 1 year
  mobility (0 = None; 1 = Present) at 4 months and 1 year
postoperative morbidities H | 4 months, 1 year
  neuropathies (0 = None; 1 = Present) at 4 months and 1 year
postoperative morbidities I | 4 months, 1 year
  paresthesia (0 = None; 1 = Present) at 4 months and 1 year
postoperative morbidities J | 4 months, 1 year
  radiolucent lesion (0 = None; 1 = Present) at 4 months and 1 year
postoperative morbidities C | 1 week, 4 months, 1 year
  semi-quantitative assessment of swelling (0 = No swelling, 1 = Mild swelling, 2 = Moderate swelling, 3 = Severe swelling)
postoperative morbidities D | 1 week, 4 months, 1 year
  semi-quantitative assessment of ecchymosis (0 = None; 1 = Present)
survival rate | 4 months, 1 year
  presence or absence of implant (% survival)
probing depth | 4 months, 1 year
  probing depth in mm of peri-implant tissues around each implant
modified plaque index | 1 week, 4 months, 1 year
  semi-quantitative assessment of plaque around each implant(1 = Plaque only detected by running a probe along the smooth surface of the healing abutment, 2 = Plaque can be seen by the naked eye, 3 = Abundance of soft matter)
bleeding index | 4 months, 1 year
  presence or absence of bleeding after probing around each implant
suppuration | 4 months, 1 year
  presence or absence of pus exudate after probing around each implant
anxiety | preop and 1 week
  visual analog scale assessment of preoperative and postoperative anxiety (10-cm line, 0 = no anxiety, 10 = maximum anxiety)
postoperative analgesics taken | daily for 1 week
  number of analgesics taken daily after surgery
duration of surgery (minutes) | immediately postoperatively
  surgical parameters
surgical parameter | immediately postoperatively
  incision length (mm)
surgical parameter | immediately postoperatively
  implant dimensions (diameter + length in mm)
insertion torque (Ncm) | immediately postoperatively
  surgical parameter
surgical parameter | immediately postoperatively
  bone quality (Type I, II, III, IV (Lekholm & Zarb classification)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Durand, DMD, MS, Principal Investigator — Université de Montréal; Intissar Abbaoui, DDS, Study Director — Université de Montréal
Locations (1):
- Université de Montréal - Faculty of Dentistry - Dental clinics, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adell R. Tissue integrated prostheses in clinical dentistry. Int Dent J. 1985 Dec;35(4):259-65. PMID 3912327
- [Background] Ireland RS, Palmer NO, Lindenmeyer A, Mills N. An investigation of antibiotic prophylaxis in implant practice in the UK. Br Dent J. 2012 Oct;213(8):E14. doi: 10.1038/sj.bdj.2012.960. PMID 23099724
- [Background] Deeb GR, Soung GY, Best AM, Laskin DM. Antibiotic Prescribing Habits of Oral and Maxillofacial Surgeons in Conjunction With Routine Dental Implant Placement. J Oral Maxillofac Surg. 2015 Oct;73(10):1926-31. doi: 10.1016/j.joms.2015.05.024. Epub 2015 Jun 6. PMID 26101074
- [Background] Braun RS, Chambrone L, Khouly I. Prophylactic antibiotic regimens in dental implant failure: A systematic review and meta-analysis. J Am Dent Assoc. 2019 Jun;150(6):e61-e91. doi: 10.1016/j.adaj.2018.10.015. Epub 2019 Apr 20. PMID 31010572
- [Background] Esposito M, Grusovin MG, Worthington HV. Interventions for replacing missing teeth: antibiotics at dental implant placement to prevent complications. Cochrane Database Syst Rev. 2013 Jul 31;2013(7):CD004152. doi: 10.1002/14651858.CD004152.pub4. PMID 23904048
- [Background] Macy E, Contreras R. Health care use and serious infection prevalence associated with penicillin "allergy" in hospitalized patients: A cohort study. J Allergy Clin Immunol. 2014 Mar;133(3):790-6. doi: 10.1016/j.jaci.2013.09.021. Epub 2013 Nov 1. PMID 24188976
- [Background] Miller RS, Wongsrichanalai C, Buathong N, McDaniel P, Walsh DS, Knirsch C, Ohrt C. Effective treatment of uncomplicated Plasmodium falciparum malaria with azithromycin-quinine combinations: a randomized, dose-ranging study. Am J Trop Med Hyg. 2006 Mar;74(3):401-6. PMID 16525097
- [Background] Noedl H, Krudsood S, Chalermratana K, Silachamroon U, Leowattana W, Tangpukdee N, Looareesuwan S, Miller RS, Fukuda M, Jongsakul K, Sriwichai S, Rowan J, Bhattacharyya H, Ohrt C, Knirsch C. Azithromycin combination therapy with artesunate or quinine for the treatment of uncomplicated Plasmodium falciparum malaria in adults: a randomized, phase 2 clinical trial in Thailand. Clin Infect Dis. 2006 Nov 15;43(10):1264-71. doi: 10.1086/508175. Epub 2006 Oct 12. PMID 17051490
- [Background] Gomi K, Yashima A, Iino F, Kanazashi M, Nagano T, Shibukawa N, Ohshima T, Maeda N, Arai T. Drug concentration in inflamed periodontal tissues after systemically administered azithromycin. J Periodontol. 2007 May;78(5):918-23. doi: 10.1902/jop.2007.060246. PMID 17470027
- [Background] Haffajee AD, Torresyap G, Socransky SS. Clinical changes following four different periodontal therapies for the treatment of chronic periodontitis: 1-year results. J Clin Periodontol. 2007 Mar;34(3):243-53. doi: 10.1111/j.1600-051X.2006.01040.x. PMID 17309596
- [Background] Giamarellos-Bourboulis EJ. Macrolides beyond the conventional antimicrobials: a class of potent immunomodulators. Int J Antimicrob Agents. 2008 Jan;31(1):12-20. doi: 10.1016/j.ijantimicag.2007.08.001. Epub 2007 Nov 1. PMID 17935949
- [Background] Tamaoki J, Kadota J, Takizawa H. Clinical implications of the immunomodulatory effects of macrolides. Am J Med. 2004 Nov 8;117 Suppl 9A:5S-11S. doi: 10.1016/j.amjmed.2004.07.023. PMID 15586558